CLINICAL TRIAL: NCT02949505
Title: Impact of Exercise Therapy on Functional Capacity in Patients Listed for Liver Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Matthew Armstrong (Other)
Collaborators: Queen Elizabeth Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor-Investigator, Matthew Armstrong, Principal investigator, Specialist Registrar in Hepatology and Honorary Clinical Fellow, University of Birmingham
Organization: University of Birmingham (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QEUHB001
Record Dates: First submitted 2016-10-25; First posted 2016-10-31 (Estimated); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Liver Cirrhosis; Liver Dysfunction
Keywords: Prehabilitation; liver transplant; functional capacity; exercise
MeSH Terms: conditions — Liver Cirrhosis; Liver Diseases; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Experimental): 12-week home prehabilitation program
  Interventions: Behavioral: Home prehabilitation program

INTERVENTIONS:
Behavioral: Home prehabilitation program — 12-week exercise therapy using daily step program (accelerometer), functional resistance exercise sessions and telephone/virtual clinic appointments

SUMMARY:
A UK prospective, single-centre feasibility study investigating the effects of exercise therapy on functional capacity in patients on the waiting list for liver transplantation. Patients will receive a 12-week home prehabilitation program (daily step program; functional resistance exercise sessions; telephone health call or virtual clinic). The following will be assessed at weeks 0, 6 and 12 weeks: feasibility (recruitment, compliance, safety, patients perception), functional capacity (ISWT, SPBT), psychological wellbeing (HADS questionnaire) and quality of life (EQ-5D)

DETAILED DESCRIPTION:
as above

ELIGIBILITY:
Inclusion Criteria:

* Meet the United Kingdom Liver Transplant criteria for listing
* Accepted on the liver transplant waiting list for a primary transplant
* Adults ≥18years who have an indication for a liver transplant
* Diagnosed with sarcopenia at liver transplant assessment

Exclusion Criteria:

* Significant cardiovascular instability including a recent Myocardial infarction, recent Cerebrovascular accident and/or a recent unstable arrhythmia
* Unstable encephalopathy - open to interpretation by the chief investigator
* Patient or next of kin non-English speaking
* Inpatients
* Refusal or lacks capacity to give informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with intervention-related adverse events as assessed by CTCAE v4.0 | 12-week
  As this is a feasibility/Pilot study the investigators need to assess if any participants have any adverse events related to the home prehabilitation programme and if so, determine the severity and frequency

OTHER OUTCOMES:
Functional capacity - incremental shuttle walk test | 12-weeks
  incremental shuttle walk test
Functional capacity - short performance battery test | 12-weeks
Psychological wellbeing - HADS questionnaire | 12-weeks
  HADS questionnaire
Quality of Life - EQ-5D questionnaire | 12-weeks
  EQ-5D questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: James Ferguson, phD, Principal Investigator — Queen Elizabeth University Hospital Birmingham; Felicity Williams, Principal Investigator — Queen Elizabeth University Hospital Birmingham
Locations (1):
- Queen Elizabeth University Hospital Birmingham, Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Williams FR, Vallance A, Faulkner T, Towey J, Kyte D, Durman S, Johnson J, Holt A, Perera MT, Ferguson J, Armstrong MJ. Home-based exercise therapy in patients awaiting liver transplantation: protocol for an observational feasibility trial. BMJ Open. 2018 Jan 21;8(1):e019298. doi: 10.1136/bmjopen-2017-019298. PMID 29358444